CLINICAL TRIAL: NCT05126992
Title: A Post-authorisation/Post-marketing Observational Study to Evaluate the Association Between Exposure to AZD1222 and Safety Concerns Using Existing Secondary Health Data Sources
Brief Title: EU Secondary Data Post-Authorisation Safety Study of AZD1222
Acronym: D8111R00006
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: D8111R00006
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: COVID-19, Vaccine Adverse Events of Special Interest
Keywords: AZD1222; ChAdOx1nCoV-19; Vaccine Adverse Events of Special Interest
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AZD1222: at least one dose of AZD1222
  Interventions: Biological: AZD1222
- comparator 1: concurrent unvaccinated
- comparator 2: historical controls
- comparator 3: active comparators*
  *Feasibility of the active comparator analysis will be assessed prior to conducting the analysis to ensure comparability between groups

INTERVENTIONS:
Biological: AZD1222 — Covid-19 AstraZeneca Vaccine
  Groups: AZD1222

SUMMARY:
A study based on electronic heath records will evaluate the incidence and relative risk of safety concerns and adverse events of special interest (AESIs) following immunisation by AZD1222 in the real-world setting.

A cohort and a self-controlled case series desings will be used.

DETAILED DESCRIPTION:
This retrospective study based on electronic heath records will evaluate the incidence and relative risk of safety concerns and adverse events of special interest (AESIs) following immunisation by AZD1222 in the real-world setting. The primary study objectives are to (1) describe baseline characteristics of all individuals in the matched population over the study period; (2) describe, among subjects who receive a first dose of AZD1222, the timing and type of second dose of any COVID-19 vaccine over the study period; (3) describe the incidence of prespecified AESIs in subjects who have received at least one dose of AZD1222 in the matched population and unvaccinated subjects; and (4) estimate any increased risk of prespecified AESIs following vaccination with AZD1222 using study retrospective cohort and self-controlled risk interval designs. Secondary objectives are identical to the primary, although focused on specific populations considered to have missing information, specifically (a) women who are pregnant or breastfeeding, (b) immunocompromised patients, (b) frail patients with certain comorbidities, (c) patients with autoimmune or inflammatory disorders, and (d) patients who, at cohort entry, had recently received a number of selected vaccines to prevent diseases other than COVID-19. A cohort and a self-controlled case series designs will be used.

Exploratory objectives: 1) To describe the IRs of prespecified AESIs in subjects who received an mRNA vaccine against COVID-19 (either Comirnaty or Spikevax) (active comparators) and in subjects from the pre-pandemic period (2017-2018) (historical comparators) in the matched population; 2) To estimate the relative and absolute risk of prespecified AESIs in subjects who received at least 1 dose of AZD1222 in the matched population compared with historical comparators in the matched population; and 3) To estimate the relative and absolute risk of prespecified AESIs in subjects who received 2 doses of AZD1222 in the matched population compared with subjects who received 2 doses of active comparator (Comirnaty or Spikevax as per homologous vaccination regimen) in the matched population*

*Feasibility of the active comparator analysis will be assessed prior to conducting the analysis to ensure comparability between groups.

ELIGIBILITY:
Inclusion criteria for AZD1222, unvaccinated, and active comparators*:

* Have at least 12 months of data available before the index date
* Have no record of vaccination with any other COVID-19 vaccine on or before the index date

Inclusion criteria for historical comparators:

- Have at least 12 months of data available before the index date

Exclusion criteria:

For each AESI, subjects (in any matched cohort) who had a specific AESI during the look-back period before the index date will be excluded from the cohort for the analysis of that specific AESI, but not from the cohorts for analysis of other AESIs.

- If a subject had a specific AESI between the index date and the start of the risk window or had any censoring criteria within this time period, the subject will be excluded from the analysis of that specific AESI.

*Feasibility of the active comparator analysis will be assessed prior to conducting the analysis to ensure comparability between groups

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include subjects who are exposed to the AZD1222 vaccine and 3 comparator groups: concurrent subjects who have not received any SARS-CoV-2 vaccine, historical controls, and active comparators*
  *Feasibility of the active comparator analysis will be assessed prior to conducting the analysis to ensure comparability between groups
Sampling Method: Non-Probability Sample
Enrollment: 5321930 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Adverse events of special interest | up to 365 days
  several AESIs

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Rebordosa, MD, PhD, Principal Investigator — RTI
Locations (4):
- Research Site, Utrecht, Netherlands
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Valencia
- Research Site, Southampton, United Kingdom

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111R00006&attachmentIdentifier=476d25e9-adb1-4e10-87ea-dd5db181b405&fileName=D8111R00006_CSR_Synopsis.pdf&versionIdentifier=